CLINICAL TRIAL: NCT00152178
Title: The Comparative Trial of UFT + TAM With CMF + TAM in Adjuvant Therapy for Breast Cancer (CUBC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91023033
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tegafur; Uracil; Tamoxifen; Methotrexate; Fluorouracil

ARMS (2):
- 1 (Experimental): UFT (uracil, tegafur) and tamoxifen
  Interventions: Drug: UFT (uracil, tegafur) and tamoxifen
- 2 (Active Comparator): CMF(cyclophosphamide, methotrexate, fluorouracil) and tamoxifen
  Interventions: Drug: CMF(cyclophosphamide, methotrexate, fluorouracil) and tamoxifen

INTERVENTIONS:
Drug: UFT (uracil, tegafur) and tamoxifen — UFT(uracil, tegafur:270 mg/m2/day (p.o.) for 2 years) and tamoxifen:20 mg/body/day(p.o.) for 2 years.
  Arms: 1
Drug: CMF(cyclophosphamide, methotrexate, fluorouracil) and tamoxifen — CMF 6 cycles(q28 days X 6 cycles of cyclophosphamide:65mg/m2/day(p.o.)day 1-14, methotrexate:40mg/m2(i.v.)day 1,8 and fluorouracil:500mg/m2(i.v.)day 1,8) and tamoxifen:20mg /body/day(p.o.) for 2 years.
  Arms: 2

SUMMARY:
This controlled study is designed to evaluate the relapse-free survival of UFT + TAM compared with CMF + TAM. Patients are randomly assigned to receive either CMF + TAM or UFT + TAM within 6 weeks after surgery. To assess treatment efficacy, data on recurrence and survival will be collected for 5 years after surgery. To evaluate the safety, data on adverse events will be collected during treatment. Patients'quality of life will be assessed by means of a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 65
* Hematopoietic WBC ≥ 4,000/mm^3 Platelet ≥ 100,000/mm^3 Hemoglobin ≥ 11.0 g/dL
* Hepatic AST and ALT ≤ 40 U/L Total bilirubin ≤ 1.5 mg/dL
* Renal BUN ≤ 25 mg/dL Creatinine ≤ 1.5 mg/dL

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 1996-07; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival | recurrence and survival will be collected for 5 years after surgery

SECONDARY OUTCOMES:
Overall survival, adverse events, and the quality of life | adverse events will be collected during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Koyama, MD, Principal Investigator — Osaka Medical Center for Cancer and Cardiovascular Diseases
Locations (1):
- Osaka Medical Center for Cancer and Cardiovascular Diseases, 1-1-3, Nakamichi, Higashinari-ku, Osaka, Osaka, Japan

REFERENCES:
- [Result] Park Y, Okamura K, Mitsuyama S, Saito T, Koh J, Kyono S, Higaki K, Ogita M, Asaga T, Inaji H, Komichi H, Kohno N, Yamazaki K, Tanaka F, Ito T, Nishikawa H, Osaki A, Koyama H, Suzuki T. Uracil-tegafur and tamoxifen vs cyclophosphamide, methotrexate, fluorouracil, and tamoxifen in post-operative adjuvant therapy for stage I, II, or IIIA lymph node-positive breast cancer: a comparative study. Br J Cancer. 2009 Aug 18;101(4):598-604. doi: 10.1038/sj.bjc.6605218. Epub 2009 Jul 28. PMID 19638976